CLINICAL TRIAL: NCT03237455
Title: Magnetic Resonance Imaging in High Risk Patients for the Development of Diffuse Idiopathic Skeletal Hyperostosis (DISH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Reuven Mader, Associate clinical professor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0102-17-EMC
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hyperostosis, Diffuse Idiopathic Skeletal; Metabolic Syndrome; Diabetes Mellitus
MeSH Terms: conditions — Hyperostosis, Diffuse Idiopathic Skeletal; Metabolic Syndrome; Diabetes Mellitus | interventions — Diagnostic Imaging; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: case control study
Who Masked: Outcomes Assessor
Masking Description: Reader of the MRI studies will be blinded to the patients diagnoses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Thoracic spine x-rays+whole spine MRI blood tests constitutional and demographic data collection
  Interventions: Diagnostic Test: Thoracic spine x-rays+whole spine MRI; Diagnostic Test: blood tests; Other: constitutional and demographic data collection
- control group (Active Comparator): Thoracic spine x-rays+whole spine MRI blood tests constitutional and demographic data collection
  Interventions: Diagnostic Test: Thoracic spine x-rays+whole spine MRI; Diagnostic Test: blood tests; Other: constitutional and demographic data collection

INTERVENTIONS:
Diagnostic Test: Thoracic spine x-rays+whole spine MRI — PA radiographs of the thoracic spine and MRI of the whole spine and sacroiliac joints
  Other Names: imaging
Diagnostic Test: blood tests — blood chemistry including total cholesterol, LDL HDL, CBC, HbA1C, fasting glucose, TG, and insulin levels, HLA-B27, 2 vials of frozen serum for future studies.
  Other Names: laboratory
Other: constitutional and demographic data collection — demographics, concomitant diseases (in particular type 2 DM, hypertension, hyperlipidemia) concomitant medications, height and weight (BMI), waist circumference
  Other Names: data

SUMMARY:
Diffuse idiopathic skeletal hyperostosis (DISH) is a poorly understood, systemic condition characterized by progressive calcification and ossification of ligaments and entheses. The current classification criteria allow diagnosing the disease in its late course, when significant bony overgrowth already involves the vertebral column and the appendicular skeleton. The research of the pathogenic mechanisms in DISH, is significantly hampered by the late diagnosis resulting from this definition.Based on recent MRI studies in both axial spondyloarthritis (axSpA) and in DISH, it seems that changes similar to the classical early inflammatory changes described in axSpA, can be detected in patients with DISH. We therefore hypothesize, that patients with metabolic syndrome without radiographic evidence for spinal DISH, might exhibit early MRI changes. If this hypothesis proves to be correct, early diagnosis and research of the possible pathogenetic mechanisms at this early stage might be very rewarding in investigations of the early aberrations of the entheses homeostasis and eventually early, more targeted therapeutic interventions. The study will examine MRI changes in patients, in their 5th decade of life, with high risk for the development of DISH (ie diabetes mellitus, metabolic syndrome) compared with patients who don't have this risk.

DETAILED DESCRIPTION:
Patient's selection- Patients will be recruited from obesity/metabolic/diabetes clinics and from bariatric surgeries clinics. All patients will have the diagnosis of metabolic syndrome National Cholesterol Education Panel III (NCEP). Patients in their 5th decade of life will be recruited for the study. This study group will have to meet the NCEP 3 criteria for metabolic syndrome and/or have type 2 diabetes mellitus (9). An age and sex matched individuals who do not meet these pre-requisits will serve as a control group.

All asymptomatic patients will undergo postero-anterior and lateral x-rays of the thoracic spine, unless they have postero-anterior or lateral thoracic spine or chest x-rays in the year preceding the recruitment. For patients with back pain, addition of cervical or lumbar spine radiographs will be permitted based on the physician judgement. Patients recruited for the study will have a total spine and sacroiliac MRI (see below) read by radiologists and rheumatologists, expert in musculoskeletal imaging, who will be blinded for the patient's data. The readings of the radiographs and the MRI will be performed in a random order.

All patients and controls will undergo postero anterior and lateral thoracic spine X-rays and MRI of the entire spine and their sacroiliac joints (Spine: sagittal T1-weighted and T2 with fat suppression sequences, SIJ semicoronal T1-weighted and T2 with fat suppression sequences) at study entry.

An accepted scoring system for the interpretation of the MRI studies will be employed for both the spine and the sacroiliac joints.

ELIGIBILITY:
Inclusion Criteria:

* Meet the NCEP 3 criteria for metabolic syndrome and/or have type 2 diabetes mellitus (9).

Age 40-49 years

Exclusion Criteria:

* ESR and CRP levels above common levels adjusted for age, gender, and weight.(I have ref for the determination of common CRP levels).

Positive HLA B-27 Personal or family history of Spondyloarthritis, psoriasis or inflammatory arthritis (past or present) Inflammatory back pain as defined by the ASAS definition (age at onset <40y, insidious onset, improvement with exercise, no improvement with rest, pain at night with improvement upon getting up = IBP if 4/5 items are present) (Ref) History of uveitis Plain radiographs with evidence for DISH

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory changes in the spine and/or sacroiliac joints | 6 months
  inflammatory bone marrow edema lesions and fatty lesions and the anterior and posterior corners of the spine (Berlin score) as well as for the presence of enthesitis on the posterior elements.
  The sacroiliac joints will also be scored according to the Berlin scoring method for the presence of acute and structural inflammatory lesion, including BME, fat metaplasia, erosions, sclerosis, ankylosis. Anterior and posterior extraarticular enthesitis will also be registered

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Mader, MD, Principal Investigator — HaEmek MC
Locations (1):
- HaEmek MC and Chaim Sheba MC, Afula, Israel

IPD SHARING:
Plan to Share IPD: No
Other researchers are expected to perform the study in their own countries. If they perform the study, unidentified data from the present study will be processed with the other parties data.

REFERENCES:
- [Background] Mader R, Verlaan JJ, Buskila D. Diffuse idiopathic skeletal hyperostosis: clinical features and pathogenic mechanisms. Nat Rev Rheumatol. 2013 Dec;9(12):741-50. doi: 10.1038/nrrheum.2013.165. Epub 2013 Nov 5. PMID 24189840
- [Background] Mader R, Novofestovski I, Adawi M, Lavi I. Metabolic syndrome and cardiovascular risk in patients with diffuse idiopathic skeletal hyperostosis. Semin Arthritis Rheum. 2009 Apr;38(5):361-5. doi: 10.1016/j.semarthrit.2008.01.010. Epub 2008 Mar 4. PMID 18304611
- [Background] Mader R, Buskila D, Verlaan JJ, Atzeni F, Olivieri I, Pappone N, Di Girolamo C, Sarzi-Puttini P. Developing new classification criteria for diffuse idiopathic skeletal hyperostosis: back to square one. Rheumatology (Oxford). 2013 Feb;52(2):326-30. doi: 10.1093/rheumatology/kes257. Epub 2012 Sep 29. PMID 23024057
- [Background] Weiss BG, Bachmann LM, Pfirrmann CW, Kissling RO, Zubler V. Whole Body Magnetic Resonance Imaging Features in Diffuse Idiopathic Skeletal Hyperostosis in Conjunction with Clinical Variables to Whole Body MRI and Clinical Variables in Ankylosing Spondylitis. J Rheumatol. 2016 Feb;43(2):335-42. doi: 10.3899/jrheum.150162. Epub 2015 Dec 15. PMID 26669910
- [Background] Mader R, Novofastovski I, Iervolino S, Pavlov A, Chervinsky L, Schwartz N, Pappone N. Ultrasonography of peripheral entheses in the diagnosis and understanding of diffuse idiopathic skeletal hyperostosis (DISH). Rheumatol Int. 2015 Mar;35(3):493-7. doi: 10.1007/s00296-014-3190-0. Epub 2014 Dec 13. PMID 25503650
- [Background] Arad U, Elkayam O, Eshed I. Magnetic resonance imaging in diffuse idiopathic skeletal hyperostosis: similarities to axial spondyloarthritis. Clin Rheumatol. 2017 Jul;36(7):1545-1549. doi: 10.1007/s10067-017-3617-6. Epub 2017 Mar 31. PMID 28364275
- [Background] Julkunen H, Heinonen OP, Pyorala K. Hyperostosis of the spine in an adult population. Its relation to hyperglycaemia and obesity. Ann Rheum Dis. 1971 Nov;30(6):605-12. doi: 10.1136/ard.30.6.605. No abstract available. PMID 5130140
- [Background] 8. Mader R, Fawaz A, Bieber A, Novofastovski I. Diffuse idiopathic skeletal hyperostosis (DISH) of young adults: lessons to be learnt. Austin J Orthopade & Rheumatol. 2016; 3(4): 1043.
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Landewe RB, Hermann KG, van der Heijde DM, Baraliakos X, Jurik AG, Lambert RG, Ostergaard M, Rudwaleit M, Salonen DC, Braun J. Scoring sacroiliac joints by magnetic resonance imaging. A multiple-reader reliability experiment. J Rheumatol. 2005 Oct;32(10):2050-5. PMID 16206369